CLINICAL TRIAL: NCT06552039
Title: Scientific Evaluation of the Safety and Efficacy of Herbal and Non Herbal Formulations in Mitigating Hair Fall, Promoting Hair Growth, and Preventing Premature Hair Graying.
Brief Title: Proof-of-Science, Prospective, Interventional, Three-arm, Double-Blind, Randomized, Safety and Efficacy Real World Evidence Study.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NovoBliss Research Pvt Ltd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: NB230043-NB
Record Dates: First submitted 2024-07-30; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Hair Fall and Pre-mature Graying

STUDY DESIGN:
Intervention Model Description: Proof-of-Science, Prospective, Interventional, Three-arm, Double-Blind, Randomized, Safety and Efficacy
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Polyherbal Hair Oil (Experimental): Apply oil with the help of fingertips on your scalp and massage it gently enabling it to penetrate into the roots (follicle) of your hair. Don't apply with your palms and never rub it vigorously as it may uproot weak hair. Let the oil gradually seep into follicle of your hair & nourish them for the whole night. The oil may be removed in the morning by washing of hair with Ayurvedic Shampoo.
  Dosage form: Liquid Frequency: Three times a week Route of Administration: Topical
  Interventions: Other: Polyherbal Hair Oil
- Minoxidil Herbal Hair Oil + Minoxidil 5 (%) Hair Serum (Active Comparator): First, apply the herbal hair oil generously to your scalp and hair, ensuring thorough coverage. Gently massage it in with your fingertips to promote circulation and absorption. After the oil application, follow the instructions provided for the application of the minoxidil hair serum. Apply the serum to the areas of your scalp where you desire hair growth, using the dropper provided or as directed. Massage it gently into your scalp to ensure even distribution and absorption. Leave the serum on without rinsing Frequency: For Minoxidil - Daily Night Application For Herbal Hair Oil- Thrice a week Route of Administration: Topical
  Interventions: Other: Minoxidil Herbal Hair Oil + Minoxidil 5 (%) Hair Serum
- Minoxidil Hair Serum (Active Comparator): Apply the amount prescribed to the area of the scalp being treated, beginning in the center of the area. Frequency: Daily Night Application of Minoxidil Route of Administration: Topical
  Interventions: Other: Minoxidil Hair Serum

INTERVENTIONS:
Other: Polyherbal Hair Oil — Apply oil with the help of fingertips on your scalp and massage it gently enabling it to penetrate into the roots (follicle) of your hair. Don't apply with your palms and never rub it vigorously as it may uproot weak hair. Let the oil gradually seep into follicle of your hair & nourish them for the whole night. The oil may be removed in the morning by washing of hair with Ayurvedic Shampoo. Dosage form: liquid frequency: Three times a week Route of Administration: Topical
  Arms: Polyherbal Hair Oil
Other: Minoxidil Herbal Hair Oil + Minoxidil 5 (%) Hair Serum — First, apply the herbal hair oil generously to your scalp and hair, ensuring thorough coverage. Gently massage it in with your fingertips to promote circulation and absorption. After the oil application, follow the instructions provided for the application of the minoxidil hair serum. Apply the serum to the areas of your scalp where you desire hair growth, using the dropper provided or as directed. Massage it gently into your scalp to ensure even distribution and absorption. Leave the serum on without rinsing.
  Dosage form: liquid Frequency : For Minoxidil - Daily Night Application For Herbal Hair Oil- Thrice a week.
  Route of Administration: Topical
  Arms: Minoxidil Herbal Hair Oil + Minoxidil 5 (%) Hair Serum
Other: Minoxidil Hair Serum — Apply the amount prescribed to the area of the scalp being treated, beginning in the center of the area. Dosage form: liquid Frequency : Daily night Application of Minoxidil Route of Administration: Topical
  Arms: Minoxidil Hair Serum

SUMMARY:
This is proof-of-science, prospective, interventional, three-arm, double-blind, randomized, safety and efficacy real world evidence study of herbal and non herbal formulations in healthy human subjects having complaint of hair fall and pre-mature graying.

DETAILED DESCRIPTION:
Considering the clinical safety, efficacy study a sufficient number 99 subjects (33 subject/arm) will be enrolled to 90 subjects (30 subject/arm) completed the study. In each arm, fifteen (15) participants per group will be recruited, with one group consisting of individuals experiencing mild to moderate Androgenetic Alopecia (AGA) class 1, 2, 3, while the other group will comprise fifteen (15) healthy subjects with symptoms of hair loss and premature graying. The potential subjects will be screened as per the inclusion & exclusion criteria only after obtaining written informed consent from the subjects. The adult female/male subjects will be instructed to visit the facility as per the below visits.

* Visit 01 (Day -04): Screening, Tattoo creation, Hair Growth Rate measurement
* Visit 02 (Day 01): Enrolment, Hair Growth Rate measurement, All evaluations
* Visit 03 (Day 45 (±2 days)): Treatment Phase
* Visit 04 (Day 87 (±2 days)): Treatment Phase, Tattoo creation, Hair Growth Rate measurement Visit 05 (Day 90 (3 days from visit 04): Hair Growth Rate measurement, All evaluations
* Visit 06: (Day 120 (±2 days)): End of Treatment Phase, All evaluations

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 55 years and above (both inclusive) at the time of consent.
2. Sex: Males and non-pregnant/non-lactating females (preferably equal number of males and females).
3. Females of childbearing potential must have a self-reported negative urine pregnancy.
4. Subject is in good general health as determined by the Investigator on the basis of medical history.
5. Female with 40-50 counts and male with 25 -30 counts of hair fall at screening.
6. Subject having AGA and premature Gray hair at a time of screening.
7. Subject having premature gray hair at a time of screening.
8. Subject with pro-claimed nonpathological thinning of hair.
9. Subject is able to remain on stable doses of contraceptive or replacement hormonal therapy, including no therapy, 6 weeks prior to and for the duration of the study.
10. If the subject is of childbearing potential, is practicing and agrees to maintain an established method of birth control (IUD, hormonal implant device/injection, regular use of birth control pills or patch, diaphragm, condoms with spermicide or sponge with spermicidal jelly, cream or foam, partner vasectomy or abstinence). Females will beconsidered as non-childbearing potential if they are surgically sterile, have been post menopausal for at least 1 year or have had a tubal ligation.
11. Subjects are willing to give written informed consent and are willing to follow the study procedure.
12. Subjects who commit not to use any other medicated/ prescription shampoos/hair care products (containing Minoxidil), any other hair growth products or hair colour or dye, other than the test products for the entire duration of the study.
13. Willing to use test products throughout the study period.
14. Subject is willing and able to follow and allow study staff to performed study test methods.
15. Subject is willing and able to follow the study directions, to participate in the study, returning for all specified visits.
16. Subject must be able to understand and provide written informed consent to participate in the study

Exclusion Criteria:

1. Subject have history of severe hair fall due to any clinically significant problems like anaemia, thyroid problems.
2. Subject have history of any dermatological condition of the scalp other than hair loss and dandruff.
3. Subject have history of any prior hair growth procedures (e.g. hair transplant or laser).
4. Subject who had taken topical treatment of hair loss for at least 4 weeks.
5. Subject who had taken any systemic treatment for at least 3 months.
6. History of alcohol or drug addiction.
7. Subject having history or resent condition of irritated or visibly inflamed scalp or severe scalp disease.
8. Subject having history or present condition of an allergic response to any cosmetic products, any other condition which could warrant exclusion from the study.
9. Pregnant or breast feeding or planning to become pregnant during the study period.
10. History of chronic illness which may influence the cutaneous state.
11. Subject have participated any clinical research study related to hair care products.
12. Subject have history of mastectomy for cancer involving removal of lymph nodes within the past year, or treatment of any type of cancer within the last 6 months.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Estimated)
Dates: Start 2024-08-24 (Estimated); Primary Completion 2024-12-24 (Estimated); Study Completion 2024-12-24 (Estimated)

PRIMARY OUTCOMES:
change in hair thickness by using CASLite Nova | Baseline before usage of test product on Day 01 and after usage of the test products on Day 45 , Day 90 and Day 120
  To assess the effectiveness of the test products in terms of change in hair thickness by using CASLite Nova.
change in hair density by using CASLite Nova | Baseline before usage of test product on Day 01 and after usage of the test products on Day 45 , Day 90 and Day 120
  To assess the effectiveness of the test products in terms of hair density by using CASLite Nova.
change in hair growth rate by using CASLite Nova | Baseline before usage of the test products on Day 01 and after usage of the test products on Day 45 , Day 90 and Day 120 .
  To assess the effectiveness of the test products in terms of change in hair growth rate by using CASLite Nova
change in hair strength by using hair pull test. | Baseline before usage of the test products (04 days before Day 01) and after usage of the test on Day 45, Day 90 and Day 120
  To assess the effectiveness of the test products in terms of change in hair strength by using hair pull test
change in hair fall by using 60 second hair combing test. | Baseline before usage of the test products (04 days before Day 01) and after usage of the test on Day 45, Day 90 and Day 120.
  To assess the effectiveness of the test products in terms of change in hair fall by using 60 second hair combing test.
change in scalp skin hydration by using Corneometer CM 825 | Baseline before usage of the test products on Day 01 and after usage of the test products on Day 45, Day 90 and Day 120
  To assess the effectiveness of the test products in terms of change in scalp skin hydration
change in Anagen: Telogen (A: T) Ratio by using Hair Pluck Test by dermatologist. | Baseline before usage of the test products on Day 01 and after usage of the test products on Day 120
  To assess the effectiveness of the test products in terms of change in Anagen: Telogen (A: T) Ratio
change in ASFS by using ASFS scoring scale. | Baseline before usage of the test products on Day 01 and after usage of the test products on Day 45 (+2 days), Day 90 (3 days from the visit 04) and Day 120 (+2 days)
  To assess the effectiveness of the test products in terms of change in ASFS where 0-10 scale (0 means no flakes and 10 means heavy flaking)
change in GSS score by using CASLite Nova | Baseline before usage of the test products on Day 01 and after usage of the test products on Day 120 (+2 days)
  To assess the effectiveness of the test products in terms of change in GSS score

SECONDARY OUTCOMES:
change in general appearance of hair | Baseline before usage of the test products on Day 01 and after usage of the test products on Day 45, Day 90 and Day 120.
  To assess the effectiveness of the test products in terms of change in general appearance of hair where categorical variable indicated as poor, average and good scale
change in general appearance of scalp. | Baseline before usage of the test products on Day 01 and after usage of the test products on Day 45 , Day 90 and Day 120.
  To assess the effectiveness of the test products in terms of change in general appearance of scalp where categorical variable indicated none, mild, moderate and excessive
change in digital photographs of the head crown Nikon digital camera D3300 | Before usage of the test products on Day 01 and after usage of the test products on Day 45 , Day 90 and Day 120.
  To assess the effectiveness of the test products in terms of change in digital photographs of the head crown
change in products perception questionnaire by using 5-point Likert scale | Before usage of the test products on Day 01 and after usage of the test products on Day 45, Day 90 and Day 120
  To evaluate the effectiveness of the test products in terms of change in products perception questionnaire
sensorial evaluation on the hair tress by 6 expert evaluation. | Baseline and post application of the test products on Day 1 at T 60 minutes
  To assess the effectiveness of the test products in terms of sensorial evaluation on the hair tress by 6 expert evaluation
change in hair shine using glossymeter GL 200 | Baseline and post application of the test products on Day 1 at T 60 minutes
  To assess the effectiveness of the test products in terms of change in hair shine using glossymeter GL 200
change in damage repair of the hair by using SEM analysis | Baseline on Day 1 and post application of the test products at 120 Days
  To assess the effectiveness of the test products in terms of change in damage repair of the hair by using SEM analysis
change in lipid deposition of the hair by using XRF method | Baseline on Day 1 and post application of the test products at 120 Days
  To assess the effectiveness of the test products in terms of change in lipid deposition of the hair by using XRF method

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Nayan K Patel, Principal Investigator — NovoBliss Research Pvt Ltd

IPD SHARING:
Plan to Share IPD: No